CLINICAL TRIAL: NCT03052452
Title: My Nutritional Health App Testing
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of Michigan (Other); Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Brennan Spiegel, Director of Health Services Research, Cedars-Sinai Medical Center
Other Study IDs: Pro00045933
Record Dates: First submitted 2017-01-05; First posted 2017-02-14 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Gastrointestinal Irritation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: My Nutritional Health App — The My Nutritional Health app built in LifeData will be used as the data collection platform for this study. We will use the data collected in the app testing to develop population-level FAST scores.

SUMMARY:
The proposed My Nutritional Health (MNH) app is a unique tool for consumers interested in tracking their food intake and linking diet to symptoms.

The investigators will test this app for developmental purposes among a sample of 100 participants who are patients of dietitians at Cedars-Sinai Medical Center (CSMC) and the University of Michigan (UM) with varying presentation of GI symptoms and suspected food intolerances. The MNH app built on the LifeData app will be used as a data collection platform for this study and can be utilized by iOS and Android smartphone devices. The investigators will use the data collected in the app testing to develop population-level FAST scores.

The MNH app includes two integrated functions:

1. Patient Symptom and Food Consumption Reporting
2. FAST Score calculation It is important to note that, per this protocol, the MNH app will only be evaluated for developmental purposes. It is currently not meant to serve as a diagnostic tool, nor to provide referrals for patients with food and symptom patterns that may suggest a food intolerance. In this respect, our test app is not governed by FDA or other regulatory bodies, as it does not make diagnoses or offer specific guidance. The purpose of this study is only to develop normative scoring distributions of FAST within the context of patients visiting GI dietitians as part of routine care.

DETAILED DESCRIPTION:
The study aims are:

AIM 1 - To validate the FAST Instrument against existing patient-reported outcome (PRO) measures.

AIM 2 - To assess sensitivity of the FAST instrument to changes in patient diet.

Investigators will collect information about food intake and related symptoms using the MNH app to validate the FAST instrument and assess its sensitivity to change in patient diet. For this study, 100 participants who are scheduled to see participating dietitians at either Cedars-Sinai Medical Center or the University of Michigan will be recruited.

Participants will be asked to report information regarding food intake and symptoms for two weeks (one week pre- and one week post-dietitian visit). The MNH app will prompt users to log food intake and any symptoms that you are experiencing at multiple time points throughout the day. Investigators will reach out to participants via telephone during the first week of enrollment to inquire about their progress using the app, assist in troubleshooting for technical difficulties, and answer any questions.

At the end of each week, participants will be asked to respond to a standardized questionnaire about GI symptoms (the 15-item Gastrointestinal Symptom Rating Scale; GSRS) and a questionnaire about general health status (the PROMIS 10 Global Health, a 10-item questionnaire developed by NIH) through the MNH mobile app.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* New patient visit with a participating dietitian at Cedars-Sinai Medical Center or University of Michigan
* Access to modern smartphone with internet or data access, to download and use the MNH app

Exclusion Criteria:

* Pregnancy, or plan to become pregnant during study.
* Inability to understand the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from those who have made new patient appointments with participating dietitians at CSMC and University of Michigan. Patients will be recruited by email by their dietitian approximately two weeks before their scheduled appointment. If interested, they will be asked to download the LifeData app on their mobile devices and search for the My Nutritional Health app within LifeData. Once in the MNH app, participants will check for eligibility, review and complete consent forms, and answer general demographic and clinical questions. Since this study is app-based, participants must have modern smartphones with internet or data access to be eligible to participate.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Food and Symptom Tracker (FAST) Score | Daily for 2 weeks
  This scale was developed by study investigators to measure gastrointestinal symptom burden at a moment in time. Raw scores range from 0 to 210 depending on the number and severity of symptoms participants report experiencing. Scores closer to 0 indicate minimal symptom burden, while scores with higher values indicate more severe symptom burden. We will be assessing change in average FAST score pre-intervention (week 1 food and symptom logs) and post-intervention (week 2 food and symptom logs).
Change in Gastrointestinal Symptom Rating Scale (GSRS) Scores | Once per week for 2 weeks
  The Gastrointestinal Symptom Rating Scale is a validated survey used to measure symptom burden. This scale ranges from 15 to 105. Higher GSRS scores indicate more severe symptom burden. Participants will complete this survey twice throughout the study: once right before their dietitian appointment and once seven days after their visit. We will assess change in pre-intervention GSRS scores and post-intervention GSRS scores.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scores | Once per week for 2 weeks
  The PROMIS Global Health Short Form is a 10-item validated questionnaire that measures an individual's overall health. During scoring, this questionnaire is broken down into two measures (physical health and mental health) and two additional questions that should be interpreted using raw values. The raw values for both the physical and mental health sub-scores range from 0 to 20, whereas the raw values for the two self-standing questions range from 0 to 5. To properly interpret scores, questionnaire responses are scored by the PROMIS Assessment Center Scoring Service to provide t-score distributions standardized to the United States general population. Lower PROMIS Global Health scores indicate poorer overall health, while higher values indicate better overall health. We will assess change in pre-intervention PROMIS scores right before the patient's appointment with a dietitian and post-intervention PROMIS scores seven days after the appointment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States